CLINICAL TRIAL: NCT02000323
Title: Early Enteral Nutrition in Severe Acute Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Erzhen Chen, Prefessor, Ruijin Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: RJpancreatitis02; RJpancreatitis02 (Other: RJH)
Record Dates: First submitted 2013-11-05; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Pancreatitis
Keywords: pancreatitis; enteral nutrition
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early enteral nutrition (Active Comparator): Naso-gastro-jejunal tube will be set up by X-ray within 24 hours of admission.
  * The distal end of the feeding tube would be placed at the remote end of Treitz ligament, and verified by X-ray.
  * After catharsis, Standard enteral nutrition liquid regimen （Peptisorb Liquid）will be used step by step.
  * Patients are targeted to receive calories for 25 kcal/kg/day.
  Interventions: Other: early enteral nutrition
- modified early enteral nutrition (Active Comparator): Naso-gastro-jejunal tube will be set up by X-ray within 24 hours of admission.
  * The distal end of the feeding tube would be placed at the remote end of Treitz ligament, and verified by X-ray.
  * After catharsis, Only Normal Saline were given through Naso-gastro-Jejunal tube until 2 or more followed requirements were met mean arterial pressure≥65mmHg; oxygenation index≥ 300;APCHEII≤8; intra-abdominal pressure <20mmHg).Then Standard enteral nutrition liquid regimen (Peptisorb Liquid) will be used step by step.
  * Patients are targeted to receive calories for 25 kcal/kg/day.
  Interventions: Other: modified early enteral nutrition

INTERVENTIONS:
Other: early enteral nutrition — Naso-gastro-jejunal tube will be set up by X-ray within 24 hours of admission.
  The distal end of the feeding tube would be placed at the remote end of Treitz ligament, and verified by X-ray.
  • After catharsis, Standard enteral nutrition liquid regimen will be used step by step.
  Patients are targeted to receive calories for 25 kcal/kg/day.
  nutrition form: short peptide ,1 kcal/ml,target 200k kcal/day
  Arms: early enteral nutrition
Other: modified early enteral nutrition — Naso-gastro-jejunal tube will be set up by X-ray within 24 hours of admission.
  * The distal end of the feeding tube would be placed at the remote end of Treitz ligament, and verified by X-ray.
  * After catharsis, Only Normal Saline were given through nasojejunal tube until 2 or more followed requirements were meted (mean arterial pressure≥65mmHg; oxygenation index≥ 300;APCHEII≤8; intra-abdominal pressure <20mmHg).Then Standard enteral nutrition liquid regimen (Peptisorb Liquid) will be used step by step.
  * Patients are targeted to receive calories for 25 kcal/kg/day.
  Arms: modified early enteral nutrition

SUMMARY:
to compare different time points for enteral nutrition in SAP patients

DETAILED DESCRIPTION:
There is increasing evidence that indicates Early Enteral Nutrition（EEN） may be associated with improved outcome in acute pancreatitis patients. However, some SAP patients failed to EEN. The researchers of this study aim to investigate the opportunity of EEN on the clinical outcomes of SAP patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of pancreatitis: Typical pain increase in serum lipase or amylase
2. Onset of abdominal pain within <=72h before admission
3. moderate severe or severe Acute Pancreatitis according to Atlanta criteria revisited in 2012 ffff

   Exclusion Criteria:
   * 1. Pregnancy 2.tumor 3. acute onset of chronic pancreatitis
4. chronic disease of any organ （heart lung gastrointestinal renal etc.） 5. Pre-existing disease with life expectancy < 3 months 7.receive parenteral nutrition or enteral nutrition before admitting

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-09 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
mortality | 28days
  the rate of patients died

SECONDARY OUTCOMES:
operation rate | 2 months
  The rate of patients received operation for pancreatitis debridement
fulfilling enteral nutrition target（≥25Kcal/kg/day） | 7 days
  enteral nutrition target set as ≥25Kcal/kg/day

OTHER OUTCOMES:
inta-abdominal infection | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Qiang en Mao, phd, Study Director — Emergency intensive care unit of Ruijin Hospital; Wen xu, Master, Principal Investigator — doctor
Locations (1):
- Ruijin, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Ong JP, Fock KM. Nutritional support in acute pancreatitis. J Dig Dis. 2012 Sep;13(9):445-52. doi: 10.1111/j.1751-2980.2012.00611.x. PMID 22908969